CLINICAL TRIAL: NCT05831839
Title: Effectiveness of Computerized Training of Attention and Working Memory in Post COVID-19 Patients With Cognitive Complaints
Brief Title: Computerized Training of Attention and Working Memory in Post COVID-19 Patients With Cognitive Complaints
Acronym: CO-TRAINER
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Chantal Luijkx, GZ-Psychologist in training for Clinical Neuropsychologist, Erasmus Medical Center
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: NL84105.078.23
Record Dates: First submitted 2023-04-20; First posted 2023-04-26 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: COVID-19; Cognitive Impairment; Cognition Disorder; Memory Disorders; Attention Deficit; Memory Impairment; Memory Loss; Attention Impaired
Keywords: COVID-19; cognitive failure; attention; memory; cognitive training; computerized training
MeSH Terms: conditions — COVID-19; Cognitive Dysfunction; Cognition Disorders; Memory Disorders; Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Intervention Model Description: Participants of the multicentre prospective cohort study CO-FLOW (NL NL74252.078.20) suffering from persistent cognitive complaints as measured with the Cognitive Failure Questionnaire (CFQ ) of the CO-FLOW-study, a multicentre prospective cohort study, will be invited (if they have agreed to be approached for further reaerch)
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive training 1 (Other): Randomized wait-list controlled pilot trial
  Interventions: Device: RehaCom
- Cognitive training 2 (Other): Randomized wait-list controlled pilot trial
  Interventions: Device: RehaCom

INTERVENTIONS:
Device: RehaCom — computerized cognitive training

SUMMARY:
Many post COVID-19 patients suffer from cognitive deficits, even after 1 year after hospitalization. These complaints have a huge impact on psychological well-being and quality of life. In rehabilitation programs in the Netherlands, most interventions are based on physical therapy or learning how to cope with fatigue and low levels of energy. In former studies computerized training of cognition in other populations has been proven to be effective. Knowledge on the effect of computerized training on attention and working memory in patients suffering from COVID-19 is urgently needed, and may contribute to more evidence-based rehabilitation programs for these patients. Therefore the effectiveness of computerized training of attention and working memory in post COVID-19 patients with cognitive complaints will be studied in this study.

DETAILED DESCRIPTION:
Since 2019, the world has been overwhelmed by COVID-19, a respiratory infectious disease. Current evidence suggests that approximately 10%-20% of people experience symptoms of post COVID-19 condition. Many post COVID-19 victims suffer from fatigue, cognitive deficits and / or subjective cognitive complaints, even after 1 year after hospitalization. Detailed research shows deficits in attention, both in sustained and executive components. Furthermore, less capacity of working memory, inhibition deficits and lower information processing speed is frequently reported. Fatigue and cognitive impairment have been consistently reported to be some of the most common and debilitating features of post COVID-19 condition. Like fatigue, cognitive complaints are associated with anxiety and depression and have an impact on every day functioning, return to work and account for diminished health-related quality of life (HR-QoL). There are no established and effective treatments yet for these patients. In former studies computerized training in other populations has been proven to be effective. Knowledge on the effect of computerized training on attention and working memory in patients suffering from COVID-19 is urgently needed, and may contribute to more evidence-based rehabilitation programs.

Objective: The primary aim of this study is to evaluate the effect of a computerized cognitive rehabilitation program (RehaCom) in post COVID-19 patients with cognitive complaints. The secondary aim is to evaluate the effect of this computerized cognitive rehabilitation program on subjective cognitive complaints, psychological outcome measures and HR-QoL and to assess the feasibility of the program.

Study design: Randomized wait-list controlled pilot trial.

Study population: Participants of the multicentre prospective cohort study CO-FLOW (NL74252.078.20) suffering from persistent cognitive complaints after 2 years after hospitalization as measured with the Cognitive Failure Questionnaire (CFQ ) will be invited.

Intervention: Computerized cognitive training, 10 weeks, 3 times/week 15 - 30 minutes/session.

Main study parameters/endpoints: Cognitive functioning (attention and working memory) and psychological functioning (coping, anxiety, depression) and HR-QoL, using non-invasive neuropsychological tests and standardized online questionnaires. All outcomes will be assessed pre- and post-intervention and at 3 and 6 months follow-up.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: The intervention is an online cognitive rehabilitation program, 3 times a week 15 - 30 minutes per session during 10 weeks. Participants can choose what time of the day is most convenient for them to engage in the program in their home environment. They might improve their attention and working memory, and therefore may also improve quality of life.

Personal and disease characteristics are copied from patient records collected in the CO-FLOW study and additional measurements are non-invasive and minimally physically demanding.

Completion of online questionnaires, additional neuropsychological measurements and joining the intervention require a certain time investment from patients and might lead to temporary fatigue. By a maximum duration of 30 minutes per session for online questionnaires and neuropsychological tests we aim to minimize the burden for patients.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 years and older;
* patient has sufficient knowledge of Dutch language;
* CFQ> 43 at 2 year follow-up of CO-FLOW, indicating persistent cognitive complaints;
* Computer and internet-access.

Exclusion Criteria:

* A potential participant who meets any of the following criteria will be excluded from participation in this study:

  * Incapacitated patients like patients diagnosed with dementia;
  * Patients should not be involved in concurrent rehabilitation program, cognitive behavioural therapy or psychotherapy targeting cognition, anxiety and/or depression.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
General cognition | 3 months
  The Montreal Cognitive Assessment (MoCA) will be used for general cognitive screening for all patients at baseline measurement and after the intervention.
  The MoCA is designed as a rapid screening instrument for cognitive dysfunction. It assesses different cognitive domains: attention and concentration, executive functions, memory, language, visioconstructional skills, conceptual thinking, calculations, and orientation. The possible score is 30 points; a score of ≥ 26 is considered as normal, 18-25 indicates mild cognitive impairment, 10-17 moderate cognitive impairment and < 10 severe cognitive impairment.
Attention | 6-9 months
  Change in visual selective attention, processing speed and concentration is measured in all patients with the D2 test at baseline measurement, after the intervention and at 3 months follow-up. Change in visual attention, executive function (divided attention) and processing speed is measured with the Trail Making Test (TMT A & B) at baseline measurement, after the intervention and at 3 months follow up. The Stroop Test measures mental speed, executive attention and response inhibition in all participants of the study at baseline measurement, after the intervention and at 3 months follow-up.
Working memory | 6-9 months
  Working memory is measured in all patients at baseline measurement, after the intervention and at 3 months follow-up with the use of the Digit Span Forward (DSF) and Digit Span Backward (DSB) test (part of the Wechsler adult intelligence scale). It involves the oral presentation of spans of digits. The measure has both a 7-item digits forward task and a 7-item digits backward task, each one with its own individual score.
  Together with 'calculation' (also a part of the Wechsler adult intelligence scale), an index for working memory can be calculated.

SECONDARY OUTCOMES:
Subjective cognitive complaints | 6-9 months
  The Cognitive Failures Test (CFQ) is used for all participants at baseline measurement, after the intervention and at 3 months follow-up to assess the frequency with which people experience cognitive failures in everyday life, such as absent-mindedness, slips and errors of perception, memory, and motor functioning. The total score of the scale is the sum of the ratings of the 25 individual items, yielding a score from 0-100. The CFQ has 3 sub-scales: forgetfulness, distractibility, and false triggering.
Anxiety and depression | 6-9 months
  The Dutch Hospital Anxiety and Depression Scale (HADS) is used for all participants at baseline measurement, after the intervention and at 3 months follow-up as a general measure of emotional distress and contains two sub-scales: anxiety and depression. Each sub-scale consists of 7 items, which are rated on a 0 to 3 point rating scale. Sub-scale scores ≥ 8 might indicate the presence of a depressive disorder or an anxiety disorder. Reliability and validity are adequate for several clinical populations, including multiple sclerosis and acquired brain injury.
Health-related quality of life (HR-QoL) | 6-9 months
  The EQ-5D-5L is used for all participants at baseline measurement, after the intervention and at 3 months follow-up as a measurement for HR-QoL. The EQ-5D-5L consists of the 5-item EQ-5D index (mobility, self-care, usual activities, pain/discomfort and anxiety/depression) and a visual analogue scale (EQ VAS). Psychometric properties of the Dutch version showed to be good. The five EQ-5D index items are summarized into one weighted overall score, which runs from 0 for the value of death to 1.00 for full health. The EQ VAS ranges from 0 to 100 (worst to best imaginable health state). For the general Dutch population average EQ-5D index = 0.843 and average EQ VAS = 81.36.
Fatigue | 6-9 months
  The Fatigue Assessment Scale (FAS) is used for all participants at baseline measurement, after the intervention and at 3 months follow-up as a measurement for fatigue. The FAS is a simple and short self-administered questionnaire to assess chronic fatigue. Patients' agreement with 10 statements is rated on a 5 points Likert-scale, ranging from 1 ("never") to 5 ("always"). Total scores can range from 10, indicating the lowest level of fatigue, to 50, denoting the highest.
Coping | 1 month
  The Coping Inventory for Stressful Situations (CISS-Short Form) is used at baseline measurement to measure coping styles of all participants.
  The short version of the CISS is used as a measure of coping with stressful situations. It has 21 items which are rated on a 1 to 5 point rating scale. It contains 3 subscales: task-oriented, emotion-oriented, and avoidance-oriented coping.
Personality traits neuroticism and extraversion | 1 month
  The Eysenck Personality Questionnaire Brief Version (EPQ-BV) is used at baseline measurement to measure level of neuroticism and level of extraversion of all participants.
  The EPQ-BV is a revised version of the EPQ-S to measure individuals on two primary personality traits in Eysenck's personality theory (1990). It consists of two measures, one for extraversion (12 items) and one for neuroticism (12 items).

CONTACTS AND LOCATIONS:
Overall Officials: Gerard Ribbers, Professor, Study Chair — Professor Rehabilitation Medicine and chair of the department
Locations (1):
- Rijndam Rehabilitation, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No